CLINICAL TRIAL: NCT06387121
Title: Efficacy and Safety of Low-dose Chemotherapy Combined With Immuno-targeted Drugs in Newly Diagnosed Adult Patients With Ph-negative B-cell Acute Lymphocytic Leukemia: A Prospective, Single-arm Clinical Study
Brief Title: Efficacy and Safety of Low-dose Chemotherapy Plus Immuno-targeted Drugs in Newly Diagnosed Adult Ph- B-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023060
Record Dates: First submitted 2024-03-04; First posted 2024-04-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
Keywords: Philadelphia Chromosome-Negative; Acute Lymphoblastic Leukemia; Elderly Or Unfit; Immuno-targeted Drugs; Low-dose Chemotherapy; Single-arm Clinical Study
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Cyclophosphamide; Dexamethasone; venetoclax; Inotuzumab Ozogamicin; blinatumomab; Mercaptopurine; Methotrexate; Cytarabine; Prednisone; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose chemotherapy, Venetoclax combined with immuno-targeted drugs (Experimental): The cycle of induction therapy is administered with immuno-targeted drugs (including Inotuzumab ozogamicin and/or Blinatumomab), a combination of low-dose chemotherapy (including vincristine, cyclophosphamide, dexamethasone, methotrexate and cytarabine) and Venetoclax (VEN).
  Interventions: Drug: Vincristine; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Venetoclax; Drug: Inotuzumab ozogamicin; Drug: Blinatumomab; Drug: 6-mercaptopurine; Drug: Methotrexate; Drug: Cytarabine; Drug: Prednisone
- low-dose chemotherapy combined with Venetoclax (Experimental): The cycle of induction therapy is administered with a combination of low-dose chemotherapy and VEN.
  Interventions: Drug: Vincristine; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Venetoclax; Drug: 6-mercaptopurine; Drug: Methotrexate; Drug: Cytarabine; Drug: Prednisone

INTERVENTIONS:
Drug: Vincristine — Anti-tumor alkaloids
  Other Names: VCR
Drug: Cyclophosphamide — Alkylating agent
  Other Names: CTX
Drug: Dexamethasone — Glucocorticoids
  Other Names: DEX
Drug: Venetoclax — Selective inhibitor of B-cell lymphoma 2 (Bcl-2)
  Other Names: VEN
Drug: Inotuzumab ozogamicin — A humanized monoclonal antibody-drug conjugate targeting CD22
  Other Names: INO
  Arms: low-dose chemotherapy, Venetoclax combined with immuno-targeted drugs
Drug: Blinatumomab — Bi-specific anti-CD19/CD3 antibodies
  Other Names: Blino
  Arms: low-dose chemotherapy, Venetoclax combined with immuno-targeted drugs
Drug: 6-mercaptopurine — Cell cycle-specific antitumor drug
  Other Names: 6-MP
Drug: Methotrexate — Antifolate antineoplastic drug
  Other Names: MTX
Drug: Cytarabine — Pyrimidine antimetabolites
  Other Names: Ara-C
Drug: Prednisone — Glucocorticoids
  Other Names: Pred

SUMMARY:
In the treatment of Ph-negative (Ph-) B-cell acute lymphoblastic leukemia (B-ALL) among adult patients, therapeutic outcomes remain suboptimal despite advances in chemotherapy and immunotherapy. A subset of adults with Ph- B-ALL have comorbidities or physiological limitations that preclude the safe administration of intensive regimens. In recent years, tumor immunotherapy has demonstrated promising safety and efficacy profiles in refractory or relapsed Ph- B-ALL across a wide spectrum of adult ages. These findings suggest that broader application of immunotherapy may represent a critical strategy to improve survival in this population. In this study, we propose a regimen that combines immuno-targeted agents with low-intensity chemotherapy for newly diagnosed adult patients with Ph- B-ALL. Our primary objective is to increase the rate of measurable residual disease (MRD)-negative complete remission (CR) following induction therapy, reduce the risk of relapse, and ultimately enhance overall survival.

DETAILED DESCRIPTION:
In this open-label, single-arm, Phase II study, prospective clinical trial, a total of 53 Ph-negative (Ph-) B-cell acute lymphoblastic leukemia (B-ALL) patients will be enrolled. The primary endpoint is measurable residual disease (MRD)-negative complete remission (CR) rate after induction therapy.

The first cycle of induction therapy is administered with Inotuzumab ozogamicin (INO), Venetoclax (VEN), and a combination of low-dose chemotherapy. The second cycle of induction therapy is Blinatumomab (Blino) plus VEN regimen. Alternatively, the first cycle of induction therapy is a combination of VEN and low-dose chemotherapy, and the second cycle of induction therapy is methotrexate (MTX) plus cytarabine (Ara-C) plus VEN regimen. Subsequent consolidation and maintenance therapy consist of low-dose chemotherapy, Blino, and VEN. Patients can receive chimeric antigen receptor T-Cell (CAR-T) Immunotherapy or allogeneic hematopoietic stem cell transplantation (HSCT) or receive autologous HSCT whenever possible during their first CR. Otherwise, they will finish the consolidation chemotherapy. Study patients are scheduled for follow-up for at least 5 years after the end of maintenance therapy.

The purpose of current study is to determine the efficacy and safety of low-dose chemotherapy combined with immuno-targeted drugs in newly diagnosed adult patients with Ph- B-ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed Ph-negative B-cell acute lymphoblastic leukemia according to World Health Organization (WHO) 2016 criteria
2. CD22 positive tumor cells
3. ≥18 years of age
4. Estimated survival ≥3 months
5. Consent and effective contraception for men and women of childbearing potential
6. Understanding and signing of informed consent forms and agreement to comply with study requirements.

Exclusion Criteria:

1. Burkitt lymphoma/leukemia
2. acute leukemias of ambiguous lineage
3. pregnant women
4. severe uncontrolled active infection
5. previous history of chronic liver disease (e.g. cirrhosis) or venous occlusive liver disease (VOD) or sinus obstruction syndrome (SOS)
6. History of clinically significant ventricular arrhythmia, syncope of unknown origin (not vasovagal) or sinoatrial block or higher degree atrioventricular (AV) block Chronic bradycardia state (unless permanent pacemaker implanted)
7. New or chronic hepatitis B or C infection (positive for hepatitis B surface antigen and anti-hepatitis C antibody, respectively) or known HIV seropositivity. HIV testing may need to be performed according to local regulations or practices
8. Psychiatric disorders likely to prevent the subject from completing treatment or informed consent
9. Other conditions considered unsuitable for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
MRD-negative complete remission rate measured by flow cytometry. | After induction (4 week)
  No immature cells were detected by flow cytometry when CR criteria were met after induction therapy.

SECONDARY OUTCOMES:
Complete remission (CR) rate | an expected average of 3 months
Overall survival (OS) | Up to 5 years post-registration
  From the date of registration to the date of death resulting from any cause.
Relapse free survival (RFS) | Up to 5 years post-registration
  From the date of complete remission (CR) until the date of documented relapse or death due to any cause or last follow-up.
Disease-free Survival (DFS) | Up to 5 years post-registration
  From CR1 to relapse, death from any cause or last follow-up.
Mortality | Day 30 and Day 60 of induction therapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terwilliger T, Abdul-Hay M. Acute lymphoblastic leukemia: a comprehensive review and 2017 update. Blood Cancer J. 2017 Jun 30;7(6):e577. doi: 10.1038/bcj.2017.53. PMID 28665419
- [Background] Pui CH, Yang JJ, Hunger SP, Pieters R, Schrappe M, Biondi A, Vora A, Baruchel A, Silverman LB, Schmiegelow K, Escherich G, Horibe K, Benoit YC, Izraeli S, Yeoh AE, Liang DC, Downing JR, Evans WE, Relling MV, Mullighan CG. Childhood Acute Lymphoblastic Leukemia: Progress Through Collaboration. J Clin Oncol. 2015 Sep 20;33(27):2938-48. doi: 10.1200/JCO.2014.59.1636. Epub 2015 Aug 24. PMID 26304874
- [Background] Boissel N, Auclerc MF, Lheritier V, Perel Y, Thomas X, Leblanc T, Rousselot P, Cayuela JM, Gabert J, Fegueux N, Piguet C, Huguet-Rigal F, Berthou C, Boiron JM, Pautas C, Michel G, Fiere D, Leverger G, Dombret H, Baruchel A. Should adolescents with acute lymphoblastic leukemia be treated as old children or young adults? Comparison of the French FRALLE-93 and LALA-94 trials. J Clin Oncol. 2003 Mar 1;21(5):774-80. doi: 10.1200/JCO.2003.02.053. Epub 2003 Mar 1. PMID 12610173
- [Background] O'Brien S, Thomas DA, Ravandi F, Faderl S, Pierce S, Kantarjian H. Results of the hyperfractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone regimen in elderly patients with acute lymphocytic leukemia. Cancer. 2008 Oct 15;113(8):2097-101. doi: 10.1002/cncr.23819. PMID 18720356
- [Background] Geyer MB, Hsu M, Devlin SM, Tallman MS, Douer D, Park JH. Overall survival among older US adults with ALL remains low despite modest improvement since 1980: SEER analysis. Blood. 2017 Mar 30;129(13):1878-1881. doi: 10.1182/blood-2016-11-749507. Epub 2017 Jan 25. No abstract available. PMID 28122741
- [Background] Maury S, Chevret S, Thomas X, Heim D, Leguay T, Huguet F, Chevallier P, Hunault M, Boissel N, Escoffre-Barbe M, Hess U, Vey N, Pignon JM, Braun T, Marolleau JP, Cahn JY, Chalandon Y, Lheritier V, Beldjord K, Bene MC, Ifrah N, Dombret H; for GRAALL. Rituximab in B-Lineage Adult Acute Lymphoblastic Leukemia. N Engl J Med. 2016 Sep 15;375(11):1044-53. doi: 10.1056/NEJMoa1605085. PMID 27626518
- [Background] Kantarjian H, Stein A, Gokbuget N, Fielding AK, Schuh AC, Ribera JM, Wei A, Dombret H, Foa R, Bassan R, Arslan O, Sanz MA, Bergeron J, Demirkan F, Lech-Maranda E, Rambaldi A, Thomas X, Horst HA, Bruggemann M, Klapper W, Wood BL, Fleishman A, Nagorsen D, Holland C, Zimmerman Z, Topp MS. Blinatumomab versus Chemotherapy for Advanced Acute Lymphoblastic Leukemia. N Engl J Med. 2017 Mar 2;376(9):836-847. doi: 10.1056/NEJMoa1609783. PMID 28249141